CLINICAL TRIAL: NCT04187430
Title: Validation of a Prediction Score for Recurrent C. Difficile Infection: Implementation for Treatment Algorithm Strategies
Acronym: Clostri_Score
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emilio Bouza (Other)
Collaborators: Elena Reigadas Ramirez (Unknown); Patricia Muñoz García (Unknown)
Responsible Party: Sponsor-Investigator, Emilio Bouza, Phd, MD Senior Assesor, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: MICRO.HGUGM.2019-016
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2019-12

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Retrospective Studies; Longitudinal Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective group
  Interventions: Behavioral: Retrospective
- Prospective group
  Interventions: Behavioral: Prospective

INTERVENTIONS:
Behavioral: Retrospective — Those patients with a positive sample for ICD will be randomly selected from the microbiology database.
  Groups: Retrospective group
Behavioral: Prospective — After the routine identification of a case of DCI by the microbiology laboratory, those new cases will be included in the study.
  Groups: Prospective group

SUMMARY:
The objective of the present study is to derive a high-risk R-ICD prediction rule and a prospective implementation of this prediction rule.

DETAILED DESCRIPTION:
For objectives 1 and 2, a retrospective study of the microbiology database will be carried out and the medical records will be consulted to collect the variables included in Annex 2. The other prediction rules to be compared are those of Cobo et al., Reigadas et al and Gerding et al.

We will review a total of 215 patients according to the calculation of the sample size (see section) A prospective study will also be carried out in which the positive patients for C. difficile determined by the Microbiology Service of the General University Hospital Gregorio Marañón will be included. The medical records of the selected cases will be reviewed. All patients included in the prospective study (Objective 3) will receive the information sheet and consent sheet that they must sign for this study (Annex 1). These patients will be followed and the variables included in Annex 2 will be collected.

ELIGIBILITY:
Inclusion Criteria:

* For the retrospective cohort, those patients with a positive sample for ICD will be randomly selected from the microbiology database.
* For the prospective cohort: after the routine identification of a case of DCI by the microbiology laboratory, those new cases will be included in the study.

Exclusion Criteria:

* Children under 18 years or patients with <3 faeces not trained in the last 24 hours will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Positive patients for C. difficile determined by the Microbiology Service of the General University Hospital Gregorio Marañón
Sampling Method: Probability Sample
Enrollment: 513 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Create Score | 31 december 2020
  Create a high risk of recurrence score by reviewing a retrospective cohort of patients with DCI.

CONTACTS AND LOCATIONS:
Locations (1):
- HGU Gregorio Maranon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided